CLINICAL TRIAL: NCT01974830
Title: AL1TER™: Alpha-1 Therapy, Evaluation, and Research Patient Registry
Acronym: AL1TER
Status: Completed | Type: Observational
Sponsor: Coram Clinical Trials (Other)
Responsible Party: Sponsor
Other Study IDs: CT-10-04
Record Dates: First submitted 2013-10-21; First posted 2013-11-04 (Estimated); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: Alpha-1 Anti-trypsin Deficiency
Keywords: alpha-1; anti-trypsin; pulmonary function; augmentation therayp; home care
MeSH Terms: conditions — alpha 1-Antitrypsin Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Adult Alpha-1 Patients: Adult Alpha-1 patients receiving augmentation therapy in the home through Coram

SUMMARY:
This is a longitudinal, observational, non-interventional registry study, designed to collect both retrospective and prospective real world data, on patients receiving Alpha-1 augmentation therapy in the home through Coram Specialty Infusion.The data will be collected from standard Coram homecare forms, as well as patient reported case forms.

DETAILED DESCRIPTION:
This is a longitudinal, observational, non-interventional registry study, designed to collect both retrospective and prospective data, in order to acquire real-world data on product prescribing, product use by patients, and product performance for patients receiving α1-PI therapy in a homecare and/or a Coram ambulatory infusion suite. There is no limit on the number of subjects that may participate in the registry. The AL1TER Registry will be overseen by the Principal Investigator listed on the first page of this protocol. No less than 40 physicians in the US will participate in this registry; there will be no upper limit to this number. All patients ≥18 years old, not members of a vulnerable study population, and who require α1-PI therapy may be invited to participate in this study.

Participation in the AL1TER Registry will continue as long as the subject is:

Being treated with α1-PI therapy using Coram's infusion services, Using an insurance carrier for which Coram is an approved provider, Willing to participate in this registry, and Until the Sponsor, Principal Investigator or subject decides to terminate their participation.

The data collection for this study differs from other registries in that data going into the AL1TER Registry is being collected by homecare agency personnel (i.e., pharmacists and nurses). The data will be collected from standard Coram homecare forms. AL1TER Registry data will be entered into Coram's standard patient database and processed in the same manner as for non-registry patients but will be extracted in a systematic fashion for incorporation into the AL1TER Registry. Data collected from the St. George Respiratory Questionnaire (SGRQ), and the Life Quality index Questionnaire (LQIQ), and subject medical chart review may also be entered into the AL1TER Registry database. All data will be de-identified for use when reporting results of the database.

All subjects participating in the AL1TER Registry will be informed about the Registry by the submitting investigators, or their designee. Additionally with physician permission, registry staff can contact patients via mail and phone to consent, only after patients have been accepted on Coram's service and agreed to start therapy. Collection of subject data for incorporation into the AL1TER Registry will begin only after the subject signs the informed consent form.

In addition to the standard visit/data collection already carried out by Coram, subjects will also be asked to complete two short quality of life questionnaires every six months beginning with 30 days after the date subject signs informed consent.

This registry study will continue until such time as the sponsor, Coram Clinical Trials, makes the decision to terminate data collection. At such time all submitting investigators, subjects and the IRB will be notified of study termination. Subject participation will begin from the date they sign informed consent and will continue until the sponsor, Principal Investigator, submitting investigator, or subject decides to terminate their participation or the registry itself is terminated. The authorization by a subject for use of their Protected Health Information (PHI) for the AL1TER Registry has no expiration date.

The AL1TER Registry involves compilation of the standard data collected for all patients receiving α1-PI therapy within the Coram system; data collected from the SGRQ and LQIQI, and relevant items from patient medical history, including pulmonary function tests. Since the registry is both retrospective and prospective, forms from the start of the patients care, through to the end of their care will be made available for entry into the registry, even forms that predate the signing of the ICF. Sample forms of the standard data collected for Coram patients are included in the appendices. The information that is captured for each α1-PI patient using Coram's standard forms may include:

Patient Start of Care:

Patient information (contact, date of birth, height, weight, gender, tobacco/alcohol/drug use) Age at time of development of symptoms, and age at time of diagnosis Medical/surgical history Alpha-1 Genotype Baseline FEV1 value Therapy and safety review (diagnosis, therapy, administration method, PICC length, date of insertion, etc.) Care plan

Ongoing Patient Assessment:

Patient information Changes in dosing Infections/illness Antibiotic use Primary care physician visits Emergency room visits Hospitalizations Effects from infusions Other changes in health Care plan update(s) Clinical monitoring (lab values, weight, nutrition screen, FEV1 values.)

Home Visit Assessments:

Patient information Therapy information Medical history and medications (initial and ongoing) Vital signs/weight Patient/home safety Access device for infusion therapy Nursing interventions Assessments: respiratory, cardiovascular, gastrointestinal, genitourinary, musculoskeletal, neurosensory, integumentary, endocrine, pain Medication administration information Teaching and compliance Insurance Information Insurance carriers Insurance coverage Reimbursement variances

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet the following criteria to participate in this study:

Signed informed consent Either male or female, ≥18yrs of age requiring α1-PI therapy Agree to the use of Coram's infusion services upon entry into AL1TER Registry

Exclusion Criteria:

* Patients will be excluded from participation in the study for any of the following reasons:

Currently using an insurance provider for which Coram's services are not covered/authorized Have previously participated in the AL1TER Registry and revoked consent to the use of their Protected Health Information in theAL1TER Registry database Under the age of 18, or member of a vulnerable population (prisoner, unable to understand the English version of the consent, or unable to sign consent themselves)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed with Alpha-1 anti-trypsin deficiency (any phenotype) on augmentation therapy
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2013-10; Primary Completion 2019-09-06 (Actual); Study Completion 2019-09-06 (Actual)

PRIMARY OUTCOMES:
Change in Pulmonary Function | From Baseline to 1 year
  Assessment of pulmonary function, including FEV1, at baseline and change (improvement or decline) at 1 year

SECONDARY OUTCOMES:
Change in Quality of Life | Baseline and 6 month
  Patients will self complete 2 surveys, life quality index questionnaire (LQIQ) and the St. George Respiratory questionnaire that asses patients infusion experience, health improvement of infusions, pain, and cost of infusions, as well as the improvement or decline in patients perceptions of their lung and respiratory functions and activities related to that.
Pulmonary Infections and Exacerbation | 6 months, 1 year, 2 years, 3 years.
  Number of pulmonary infections and exacerbation

CONTACTS AND LOCATIONS:
Overall Officials: Donald Schmechel, MD, Principal Investigator — Southeast Neurology and Memory Clinic
Locations (1):
- Coram Clinical Trials, Centennial, Colorado, United States